CLINICAL TRIAL: NCT01262235
Title: A Phase 1/2 Dose Escalation Study to Determine the Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous TKM-080301 in Patients With Advanced Solid Tumors
Brief Title: A Dose Finding Study of TKM-080301 Infusion in Neuroendocrine Tumors (NET) and Adrenocortical Carcinoma (ACC) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKM-PLK1-001
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cancer; Neuroendocrine Tumors; NET; Adrenocortical Carcinoma; ACC
Keywords: Solid tumor; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Neuroendocrine tumors (NET); Adrenocortical carcinoma (ACC); Carcinoid
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors; Adrenocortical Carcinoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Carcinoid Tumor | interventions — TKM-080301

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TKM-080301 (Experimental)
  Interventions: Drug: TKM-080301

INTERVENTIONS:
Drug: TKM-080301 — Repeat dose IV infusion.
  Other Names: PLK1 SNALP; TKM-PLK1

SUMMARY:
This study will be a Phase I/II, open-label, non-randomized, dose-finding trial conducted at multiple clinical centers. The study is designed to determine the safety, tolerability and PK of TKM-080301 in adult patients with solid tumors or lymphomas that are refractory to standard therapy or for whom there is no standard therapy. After the determination of the maximum tolerated dose this dose will be utilized in an expansion cohort or subjects with refractory neuroendocrine tumors (NET) or adrenocortical carcinoma (ACC) tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically and cytologically confirmed solid tumor that is refractory to standard therapy or for which no standard therapy is known to exist, or who are not candidates for standard therapy, or non-Hodgkin's lymphoma or Hodgkin's disease that is refractory to standard therapy (i.e., patients have relapsed following at least 2 prior therapies) or for which no standard therapy is known to exist. For the Neuroendocrine (NET) and adrenocortical carcinoma (ACC) expansion cohort subjects must have histologically or cytologically confirmed, measurable (per RECIST 1.1) NET or ACC tumor that is refractory to standard therapy or for which no standard therapy is known to exist, or who are not candidates for standard therapy.
* Patient has an ECOG performance status of 0 - 1,
* Patient has adequate hematologic, hepatic and renal function,
* Patient is seronegative for hepatitis B virus (HBV) and hepatitis C virus (HCV),
* Patients must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

* Unresolved toxicities (> Grade 1) of previous chemotherapy,
* Patients with primary tumors of the central nervous system (CNS),
* Prophylactic hematologic growth factors administered </= 2 weeks prior to start of therapy,
* Patient has history of or existing clinically significant cardiovascular disease,
* Patient has a history of clinically significant asthma or COPD requiring daily medication within the last 6 months,
* Patient has a seizure disorder not controlled on medication,
* Patient has a known or suspected viral, parasitic, or fungal infection,
* Patient has known hypersensitivity or previous severe reactions to oligonucleotide- or lipid-based products, including liposomal drug products and phospholipid-based products,
* Patient has been treated with any investigational drugs, biologics, or devices within 28 days prior to study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of treatment with TKM-080301 | 6 months
Determine dose-limiting toxicities and maximum tolerated dose of TKM-080301 | 6 months

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of TKM-080301 | 2 months
Assess preliminary evidence of anti-tumor activity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kowalski, MD, Study Director — Tekmira Pharmaceuticals
Locations (8):
- United States (8):
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Westchase Oncology Center, Houston, Texas